CLINICAL TRIAL: NCT00645229
Title: Efficacy And Safety Of Ziprasidone In Acute Exacerbation Of Schizophrenia Or Schizoaffective Disorder, Including Patients With A Diagnosis Of Recent Onset
Brief Title: A Study of the Efficacy and Safety of Ziprasidone in Patients With Acute Exacerbation of Schizophrenia or Schizoaffective Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281055
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Ziprasidone 20 mg capsules twice daily on Days 1-3; dose could be increased if clinically indicated up to 80 mg twice daily; total treatment duration was to be 24 weeks
  Other Names: Geodon, Zeldox

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ziprasidone in acute exacerbation of schizophrenia or schizoaffective disorder, including patients with recent onset of symptoms

DETAILED DESCRIPTION:
The study was prematurely discontinued due to the difficulty of subject recruitment on March 24, 2005. There were no safety concerns that led to the decision to terminate.

ELIGIBILITY:
Inclusion Criteria:

* Patients not currently being treated with antipsychotic medication and neuroleptic naive patients
* Diagnosis of schizophrenia or schizoaffective disorder
* Antipsychotic treatment prior to screening was to be for a cumulative period of less than 5 years

Exclusion Criteria:

* Patients at immediate risk of committing harm to self or others
* Treatment with clozapine within 3 months prior to baseline
* History of neuroleptic treatment
* Current antipsychotic treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2004-09; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) total score at Week 24 | Week 24
Change from baseline in PANSS (Depression-C) score at Week 24 | Week 24
Change from baseline in Clinical Global Impressions-Severity (CGI-S) total score at Week 24 | Week 24
Change from baseline in CGI-S total score at Week 24 | Week 24

SECONDARY OUTCOMES:
Vital signs and weight at screening, baseline, Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6 | Screening, baseline, Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6
Change from baseline in Clinical Global Impressions-Improvement (CGI-I) score at Week 24 | Week 24
Adverse events on Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6 | Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6
Change from baseline in Global Assessment of Functioning (GAF) score at Week 24 | Week 24
Laboratory parameters at screening, baseline, Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6 | Screening, baseline, Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6
Simpson-Angus Scale (SAS) at screening, baseline, Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6 | Screening, baseline, Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6
Barnes Akathisia Scale (BAS) at screening, baseline, Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6 | Screening, baseline, Day 3, Week 1, and Months 1, 2, 3, 4, 5, and 6
Electrocardiogram | Screening and Month 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Lisbon, Portugal

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281055&StudyName=A%20study%20of%20the%20efficacy%20and%20safety%20of%20ziprasidone%20in%20patients%20with%20acute%20exacerbation%20of%20schizophrenia%20or%20schizoaffective%20disorder